

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Phase II Study of Autologous Lymphocyte Infusions After Radiation Therapy to Mitigate Radiation Induced Lymphopenia and Enhance Immune Reconstitution in Patients with Solid Tumor Malignancies 2019-1164

| Subtitle: Recipient | AASSTONE CONTROL OF THE CONTROL OF T |
|---|---|
| Study Chair: Gheath Al-Atrash | |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB – a committee that reviews research studies).

#### STUDY SUMMARY

White blood cells fight infection and may kill cancer cells. Chemotherapy and radiation therapy may damage or destroy the white blood cells in your blood.

The goal of this clinical research study is to learn if collecting patients' white blood cells before standard chemotherapy and radiation and then giving them their cells after treatment can help to control the disease in patients with non-small cell lung cancer or esophageal cancer.

**This is an investigational study.** Apheresis, the procedure for collecting the white blood cells, is done using FDA-approved and commercially available methods. Receiving white blood cells after chemotherapy and radiation is investigational.

Receiving white blood cells may help prevent infections and improve your cancer treatment outcome. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You will be on active study for up to 45 days after receiving the white blood cells.

You and/or your insurance provider will be responsible for the cost of the apheresis procedure, receiving the white blood cells, and other/tests procedures performed during the study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive other investigational therapy, if available. You may choose not to have treatment for the low white blood cells count at all. The study doctor will discuss with you the possible risks and benefits of these options. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be done to help the doctor decide if you are eligible:

- Blood (about 2 teaspoons) and urine will be collected for routine testing. If you can become pregnant, part of the blood or urine samples will be used for pregnancy testing.
- You may have a chest x-ray to check the status of the disease, if you have not had a CT or CT/PET scan of the neck and chest.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

Up to 20 patients will take part in this study. All will be enrolled at MD Anderson.

## **Study Treatment**

Before you receive standard of care chemotherapy and radiation for your disease, you will have an apheresis procedure to collect white blood cells from your blood.

For this procedure, you will need to stay seated in a chair and keep both arms still for about 3 hours. During this process, your blood will flow into the machine and then directly back into your bloodstream through the second line. Blood will be drawn from 1 arm through a catheter (needle and tube) connected to the apheresis machine. Inside the machine, the white blood cells will be separated from the rest of the blood cells and collected in a sterile bag. Then, the rest of the blood cells will be returned

through a catheter to your other arm. A blood thinner called citrate will be added to the blood as it enters the machine in order to lower the risk of your blood clotting in the machine. You will sign a separate consent for the standard of care apheresis procedure.

If it is too difficult to insert the catheter for the apheresis procedure, you will be removed from the study.

After the white blood cells are collected, you will receive standard of care chemotherapy and radiation for your lung or esophageal cancer. You will sign a separate consent for these procedures.

The day after your last radiation treatment, you will receive your white blood cells by vein over about 1 hour.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

## Study Visits

### Within 30 days of study enrollment:

- You will have a physical exam.
- Blood (about 2 teaspoons) will be drawn for routine tests.
- Urine will be collected for routine tests. If you can become pregnant, part of this sample will be used for a pregnancy test. To take part in this study, you must not be pregnant.
- You will have a chest x-ray.

## On the day you have the apheresis procedure and then again before receiving your white blood cells:

- You will have a physical exam.
- Blood (about 2 teaspoons) will be drawn for routine tests and to check for viruses or bacteria that can cause diseases.
- Urine will be collected for routine tests.

## Within 3 weeks and then again 6 weeks after receiving your white blood cells:

- You will have a physical exam.
- Blood (about 4 tablespoons) will be drawn for routine tests.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

**Apheresis** may cause light-headedness, chest discomfort, nausea, vomiting, and/or fainting due to low blood pressure. The filtering process also removes platelets (the

cells that help the blood to clot). If your platelet count falls low enough, you may be at increased risk of bleeding. If this occurs, any further collection will be stopped until a blood transfusion is given.

To prevent clotting, your blood will be thinned with citrate (a blood thinner) during the apheresis procedure. Citrate decreases the calcium in the blood, sometimes causing temporary numbness and/or tingling of the fingertips and/or around the mouth. Should you experience any numbness, you must tell the nurse operating the machine. If not corrected by replacing calcium, this complication could progress to severe muscle cramps while your calcium is low.

Use of the blood-cell separator may cause air to enter the blood stream, loss of blood if the tubing should break, infection, difficulty breathing, shock, irregular heartbeat, fatigue, and/or heart failure. The needle insertion used for the apheresis procedure may cause local bruising, bleeding, and/or infection in the vein and/or on the skin around the vein.

All aspirin and ibuprofen products should be avoided at least 3 days before and also during the apheresis procedures. Any high physical activity, including contact sports such as football and basketball, should be avoided for 24 hours after the apheresis procedure.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

The **lymphocyte** (white blood cell) infusion may cause fever, chills, low blood pressure, and/or shortness of breath.

**X-rays** send a small amount of radiation though the body. All radiation adds up over a lifetime and may increase the risk of a new cancer forming.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

## **Certificate of Confidentiality**

This research is covered by a Certificate of Confidentiality (CoC) from the National Institutes of Health. The researchers with this CoC may not disclose or use information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information protected by this CoC cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below).

The CoC cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation. You should understand that a CoC does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The CoC will not be used to prevent disclosure for any purpose you have consented to.

This study may involve unpredictable risks to the participants.

## **Pregnancy Related Risks**

#### **Both Males and Females**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

#### OPTIONAL PROCEDURES FOR THE STUDY

You do not have to agree to the optional procedure in order to take part in this study. There are no benefits to you for taking part in the optional procedure. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

**Optional Procedure #1:** If you agree, before the apheresis procedure and at Weeks 3 and 6, blood (about 4 teaspoons) will be drawn to check your immune system and the number and quality of the white blood cells. You will be asked to sign separate informed consent document(s) for MD Anderson laboratory protocols LAB99-062 and/or LAB09-0307 for the blood collection.

#### **Optional Procedure Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

#### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have blood drawn to check your immune system and white blood cells?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or National Institutes of Health for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## Additional Information

4. You may ask the study chair (Dr. Gheath Al-Atrash, at 713-563-3324 any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB - a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.

5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can help you safely stop study treatment. The study doctor will also decide if you need to have any visits or tests to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, National Institutes of Health, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson. Possible reasons your participation in this study may be stopped include if the disease gets worse, if intolerable side effects occur, if you are unable to follow study directions, or if the study is stopped.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: National Institutes of Health.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

## **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and National Institutes of Health, and/or shared with other researchers and/or institutions for use in future research.

#### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples stored by National Institutes of Health may be used in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples

#### Genetic Research

Samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you.

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

## Authorization for Use and Disclosure of Protected Health Information (PHI):

A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study

results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:

- Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
- The IRB and officials of MD Anderson
- National Institutes of Health, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
- Center for International Blood and Marrow Transplantation Research (CIBMTR) and any future sponsors or licensees of the study technology
- Study monitors and auditors who verify the accuracy of the information
- Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

DATE

#### CONSENT/AUTHORIZATION

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT WITNESS TO CONSENT I was present during the explanation of the research to be performed under this protocol. SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. PRINTED NAME OF WITNESS TO THE VERBAL CONSENT. PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or her authorized representative, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation. PERSON OBTAINING CONSENT DATE PRINTED NAME OF PERSON OBTAINING CONSENT **TRANSLATOR** I have translated the above informed consent as written (without additions or subtractions) into and assisted the people (Name of Language) obtaining and providing consent by translating all questions and responses during the consent process for this participant.

 $\square$  Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line.)

NAME OF TRANSLATOR

SIGNATURE OF TRANSLATOR